CLINICAL TRIAL: NCT01498874
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Gevokizumab in Subjects With Moderate to Severe Acne Vulgaris
Brief Title: Efficacy and Safety Study of Gevokizumab to Treat Moderate to Severe Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X052120
Record Dates: First submitted 2011-12-21; First posted 2011-12-26 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Acne Vulgaris
Keywords: Acne; Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — gevokizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- low dose gevokizumab (Experimental)
  Interventions: Drug: gevokizumab
- high dose gevokizumab (Experimental)
  Interventions: Drug: gevokizumab

INTERVENTIONS:
Drug: Placebo — Sterile solution administered subcutaneously on Day 0, Day 28, and Day 56
  Arms: Placebo
Drug: gevokizumab — Sterile solution administered subcutaneously on Day 0, Day 28, and Day 56
  Arms: low dose gevokizumab
Drug: gevokizumab — Sterile solution administered subcutaneously on Day 0, Day 28, and Day 56
  Arms: high dose gevokizumab

SUMMARY:
The purpose of this study is to determine whether gevokizumab is effective in the treatment of moderate to severe acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe acne vulgaris
* Acne vulgaris unresponsive to oral antibiotics
* Willingness to maintain current habits for facial cleaning, shaving, and application of cosmetics through the end of the study

Exclusion Criteria:

* Use of medications or treatments from specified pre-treatment time periods through the end of the study
* Beard, moustache, sideburns or other facial hair that may interfere with evaluation
* Other forms of acne
* History of malignancy within 5 years
* History of allergic or anaphylactic reactions to monoclonal antibodies
* History of tuberculosis
* History of chronic systemic infections
* Female subjects who are pregnant, planning to become pregnant

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The mean absolute change from baseline in inflammatory facial lesion count at Day 84 | Baseline and Day 84

SECONDARY OUTCOMES:
The proportion of subjects with a successful treatment outcome at Day 84 | Baseline and Day 84
  Successful treatment outcome is defined as an improvement of >= 2 grades from the baseline grade on the dichotomized facial Investigator's Global Assessment scale.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Hot Springs, Arkansas
  - Riverside, California
  - San Diego, California
  - Denver, Colorado
  - New Haven, Connecticut
  - Bay City, Michigan
  - Fridley, Minnesota
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Charlotte, North Carolina
  - High Point, North Carolina
  - Raleigh, North Carolina
  - South Euclid, Ohio
  - Portland, Oregon
  - Arlington, Texas
  - Austin, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia